CLINICAL TRIAL: NCT02882503
Title: A Prospective Clinical Study of Endoscopic Ultrasound Guided Radiofrequency Ablation (EUS-RFA) for Small Benign Pancreatic Tumors
Brief Title: Endoscopic Ultrasound Guided Radiofrequency Ablation (EUS-RFA) for Small Benign Pancreatic Tumors
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201604063DIPC
Record Dates: First submitted 2016-08-24; First posted 2016-08-30 (Estimated); Last update posted 2019-07-24 (Actual); Status verified 2019-06

CONDITIONS: Neuroendocrine Tumors; Cystic Neoplasms
Keywords: Endoscopic ultrasound; Radiofrequency ablation; Pancreas
MeSH Terms: conditions — Neuroendocrine Tumors; Neoplasms, Cystic, Mucinous, and Serous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- EUS-RFA (Experimental): monopolar radiofrequency probe (1.2 mm Habib endoscopic ultrasound - radiofrequency ablation (EUS-RFA) catheter) and 19 or 22 gauge fine needle aspiration (FNA) needle
  Interventions: Device: endoscopic ultrasound - radiofrequency ablation (EUS-RFA)

INTERVENTIONS:
Device: endoscopic ultrasound - radiofrequency ablation (EUS-RFA) — Radiofrequency ablation will be applied with an innovative monopolar radiofrequency probe (1.2 mm Habib EUS-RFA catheter) placed through a 19 or 22 gauge fine needle aspiration (FNA) needle in patients with a tumor in the head of the pancreas.

SUMMARY:
Incidental pancreatic solid or cystic lesions are diagnosed with increased frequency due to the widespread use of abdominal cross-sectional imaging to investigate unrelated symptoms. Lesions such as neuroendocrine tumors (NET), mucinous cystadenomas and intraductal papillary mucinous neoplasms (IPMNs) have the potential of malignant transformation. The standard treatment of solid or cystic pancreatic lesions with malignant potential has been surgical resection, with lesions in the pancreatic head requiring a Whipple resection whereas pancreatic tail lesions are treated with distal pancreatectomy. Both types of resection carry significant morbidity and mortality. The study would like to outline the feasibility, safety, adverse events and early results of endoscopic ultrasound (EUS) - radiofrequency ablation (RFA) in pancreatic neoplasms.

DETAILED DESCRIPTION:
The intervention described was radiofrequency ablation which was applied with an innovative monopolar radiofrequency probe (1.2 mm Habib EUS-RFA catheter) placed through a 19 or 22 gauge fine needle aspiration (FNA) needle once FNA was performed in patients with a tumor in the head of the pancreas. The device had been certificated by the European Union (EU) and received Food and Drug Administration (FDA) approval in 2015. The endoscopic ultrasound (EUS) - radiofrequency ablation (RFA) is a 1 Fr wire with a working length of 190 cm, which can be inserted through the biopsy channel of a EUS. RF power is applied to the electrode at the end of the wire to coagulate tissue in the liver and pancreas. In this study, the investigators will enroll 20 patients to receiving EUS-RFA of pancreatic neoplasms with the monopolar RF probe. The follow-up period will be one year with regular monitoring. Our primary endpoint will be to evaluate pancreatic tumor ablation effect, Secondary objectives will be to evaluate the mortality and morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all of the following inclusion criteria to be eligible for this study:

  1. Cystic neoplasms in pancreatic parenchyma or outer portion of the pancreas are defined by radiologists who evaluate the images more than twice in three months. The size of benign cystic neoplasm is between 0.5-3 cm. Or surgical specialist physician considers the benign tumor that larger than 3 cm is not suitable for surgery or patients unwilling to accept surgery.
  2. Normal physical condition. Eastern Cooperative Oncology Group (ECOG) score of 0-2 and American Society of Anaesthesiologists (ASA) score ≤ 3.
  3. Normal blood coagulation. Platelet count ≥ 100 K/Μl. Prothrombin time (PT)- international normalized ratio (INR) ≦ 1.5.
  4. Prior Informed Consent Form.
  5. Life expectancy of at least 3 months.

Exclusion Criteria:

* Patients presenting with any of the following will not be enrolled into this study:

  1. Women who are pregnant or women of child-bearing potential who are not using an acceptable method of contraception.
  2. To participate in any related tumor therapy clinical trials within thirty days prior to surgery.
  3. Any active metal implanted device (eg Pacemaker)
  4. Patients who have other malignancies and have not been cured within five years.
  5. Patients with resectable pancreatic cancer.
  6. Simple pancreatic cysts (including pseudocysts) or serous cystadenoma.
  7. Cystic part of the tumor is close to blood vessels or bile duct (<0.5 cm) that might injury the related structure.
  8. Cystic pancreatic tumors originate from or associate the pancreatic ducts.
  9. Have acute pancreatitis in the past four weeks
  10. Known history of human immunodeficiency virus (HIV) infection
  11. Have cardiovascular diseases (such as acute myocardial infarction, or stroke) within the last three months
  12. Moderate to severe renal dysfunction (Estimated Glomerular Filtration Rate (eGFR) <60)
  13. Have any serious or poor control of systemic disease that are not suitable for this test and followup

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-06; Primary Completion 2019-05-07 (Estimated); Study Completion 2019-05-07 (Actual)

PRIMARY OUTCOMES:
To evaluate pancreatic tumor ablation effect | up to one year
  Using magnetic resonance cholangiopancreatography (MRCP) and/or abdominal computed tomography (CT)

SECONDARY OUTCOMES:
Symptom and adverse event monitoring | up to one year
  monitor any side effects
Physical examination | up to one year
  Complete an Eastern Cooperative Oncology Group (ECOG) evaluation
Blood Routine (CBC) | up to one year
  measure of the concentration of white blood cells, red blood cells, and platelets in the blood.
Biochemical profile | up to one year
  including CEA/CA19-9, amylase, glucose

CONTACTS AND LOCATIONS:
Overall Officials: Kai-Wen Huang, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No